CLINICAL TRIAL: NCT04577430
Title: Effects of Dexmedetomidine on Cardiac Electrophysiology in Patients Under General Anesthesia During Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20200915
Record Dates: First submitted 2020-09-19; First posted 2020-10-06 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-03

CONDITIONS: Dexmedetomidine; General Anesthesia; Cardiac Electrophysiology; Cardiac Function
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Loading dose with 0.5 μg/kg, maintenance dose with 0.5 μg/kg (Experimental): 10 min before induction of anesthesia,the loading dose of dexmedetomidine is 0.5 μg/kg, and completed in 10 minutes. The maintenance dose is 0.5 μg/kg per hour during the operation until 0.5 h before the operation finished.
  Interventions: Drug: Dexmedetomidine
- Loading dose with 1 μg/kg, maintenance dose with 0.5 μg/kg (Experimental): 10 min before induction of anesthesia,the loading dose of dexmedetomidine is 1 μg/kg, and completed in 10 minutes. The maintenance dose is 0.5 μg/kg per hour during the operation until 0.5 h before the surgery finished.
  Interventions: Drug: Dexmedetomidine
- Loading dose with 1 μg/kg, maintenance dose with 1 μg/kg (Experimental): 10 min before induction of anesthesia,the loading dose of dexmedetomidine is 1 μg/kg, and completed in 10 minutes. The maintenance dose is 1 μg/kg per hour during the operation until 0.5 h before the surgery finished.
  Interventions: Drug: Dexmedetomidine
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — The loading dose with 0.5 μg/kg, maintenance dose with 0.5 μg/kg of Dexmedetomidine is used to observe the effect on the electrophysiology of the patients' hearts
  Arms: Loading dose with 0.5 μg/kg, maintenance dose with 0.5 μg/kg
Drug: Dexmedetomidine — The loading dose with 1 μg/kg, maintenance dose with 0.5 μg/kg of Dexmedetomidine is used to observe the effect on the electrophysiology of the patients' hearts
  Arms: Loading dose with 1 μg/kg, maintenance dose with 0.5 μg/kg
Drug: Dexmedetomidine — The loading dose with 1 μg/kg, maintenance dose with 1 μg/kg of Dexmedetomidine is used to observe the effect on the electrophysiology of the patients' hearts
  Arms: Loading dose with 1 μg/kg, maintenance dose with 1 μg/kg
Drug: Normal saline — Normal saline is used to observe the effect on the electrophysiology of the patients' hearts
  Arms: Normal saline

SUMMARY:
Perioperative stress may increase the incidence of adverse events in the cardiovascular system and lead to poor prognosis. Dexmedetomidine is a highly selective α2 adrenergic receptor agonist, which can inhibit stress response and reduce hemodynamic fluctuations. In different usage plans, dexmedetomidine can have different effects on hemodynamics, myocardial electrical activity, cardiac function. The main purpose was to observe its effects on myocardial electrophysiology and cardiac function during perioperative period. The secondary purpose was to explore the optimal dose of dexmedetomidine that has the least adverse effects on perioperative electrocardia action and cardiac function

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 18 to 65
* ASA I~II
* patients undergoing elective general anesthesia
* the surgery time for 1~3 h

Exclusion Criteria:

* Preoperative ECG abnormalities, including QTc ≥440 ms (male), 460ms (female)
* abnormal cardiac conduction, prolonged QT syndrome
* heart disease history, such as pacemaker implantation, unstable angina, congestive heart failure, Heart valve disease
* antiarrhythmic drugs (β-receptor blockers, calcium channel blockers, tricyclic antidepressants, etc.) that can prolong the QT interval taken within one week before surgery
* coronary heart disease, non-sinus Heart rhythm, bradycardia, tachycardia, other arrhythmia, etc
* intraoperative HR≤45 beats/min and need drugs to increase heart rate
* previous allergy to dexmedetomidine
* preoperative electrolyte abnormalities
* emergency surgery, neurological or mental disorders , Liver and kidney dysfunction
* patients who use analgesic pumps after surgery
* refusal of patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
The length of PR,QRS,QTc,QT and Tp-e intervals and the level of iCEB | during surgery to 1 month after the surgery
  All the outcomes above should be measured at the time preparing to pump a loading dose,the time after the loading dose finished,at the end of surgery,1h after the surgery finished,24 h after the surgery finished,48 h after the surgery finished,72 h after the surgery finished,1 month after the surgery finished

SECONDARY OUTCOMES:
The level of Na+,iCa2+ | perioperative
  All the outcomes above should be measured at the time preparing to pump a loading dose,the time after the loading dose finished,1h after the beginning of the surgery,the end of surgery,1h after the surgery finished
The level of cardiac circulation efficiency | Perioperative
  All the outcomes above should be measured at the time preparing to pump a loading dose,the time after the loading dose finished,1h after the beginning of the surgery,the end of surgery,1h after the surgery finished
The level of maximum pressure gradient | Perioperative
  the time preparing to pump a loading dose,the time after the loading dose finished,the beginning of surgery, 30min after the beginning of surgery,1h after the beginning of the surgery,the end of surgery,1h after the surgery finished
The level of heart rate | Perioperative
  the time preparing to pump a loading dose,the time after the loading dose finished,the beginning of surgery, 30min after the beginning of surgery,1h after the beginning of the surgery,the end of surgery,1h after the surgery finished
The level of mean arterial blood pressure | Perioperative
The level of systemic vascular resistance | Perioperative
  the time preparing to pump a loading dose,the time after the loading dose finished,the beginning of surgery, 30min after the beginning of surgery,1h after the beginning of the surgery,the end of surgery,1h after the surgery finished
The time of eyes opening from surgery ending,the whole surgery,anesthesia | intraoperative
The dosage of propofol and remifentanil | intraoperative
Total fluid intake from entering the operating room to exiting the PACU | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Tan C, Yan S, Shen J, Wu H, Yu L, Wang Y, Tian S, Zhou W, Wu Y, Zhang Z. Effects of dexmedetomidine on cardiac electrophysiology in patients undergoing general anesthesia during perioperative period: a randomized controlled trial. BMC Anesthesiol. 2022 Aug 25;22(1):271. doi: 10.1186/s12871-022-01811-5. PMID 36008759